CLINICAL TRIAL: NCT03538392
Title: Post Market Clinical Follow-up Study - PMCF Study, Serranator® Alto
Brief Title: Serranator® Alto Post Market Clinical Follow Up (PMCF) Study
Status: Withdrawn | Type: Observational
Why Stopped: Product not available, study withdrawn
Sponsor: Cagent Vascular LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Serranator® Alto PMCF Study
Record Dates: First submitted 2018-04-24; First posted 2018-05-29 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2019-07

CONDITIONS: Peripheral Arterial Disease; Arterio-venous Fistula; Arteriovenous Graft
MeSH Terms: conditions — Peripheral Arterial Disease; Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- PAD
  Interventions: Device: Serranator® Alto
- AV Fistula
  Interventions: Device: Serranator® Alto
- AV Graft
  Interventions: Device: Serranator® Alto

INTERVENTIONS:
Device: Serranator® Alto — Serranator® Alto PTA Serration Balloon Catheter

SUMMARY:
The objective of this registry is to collect observational data under local standard of care and evaluate safety and performance of the Serranator® Alto in treatment of peripheral artery disease (PAD), or dysfunctional native or synthetic arteriovenous dialysis fistulae in a real-world scenario.

DETAILED DESCRIPTION:
Single Arm, multi-center, device registry study capturing de-identified data on a minimum of 100 subjects with peripheral artery disease (PAD) and/or dysfunctional native or synthetic arteriovenous dialysis fistulae. The study will capture acute angiographic data.

ELIGIBILITY:
* Subject requires angioplasty
* Subject has a lesion in the iliac, femoral, iliofemoral, popliteal artery, or obstructive lesion of native or synthetic arteriovenous dialysis fistulae as per the product indications for use

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of subjects with claudication or ischemic rest pain, requiring dilatation of lesions, in the iliac or femoropopliteal arteries, or dysfunctional native or synthetic arteriovenous dialysis fistulae.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Performance | The registry will collect acute procedural data through hospital discharge, no additional follow up is required. Performance data will be summarized after enrollment is complete, estimated to be 1 year.
  Device Success defined as the achievement of successful delivery, balloon inflation and deflation, and retrieval of the study device(s) with a diameter stenosis of <50% by visual assessment at the intended target site after using the Serranator® device.

SECONDARY OUTCOMES:
Collection of device related Major Adverse Events (MAE) until discharge | Within 12-24 hours post-procedure or prior to hospital discharge, whichever occurs first
  Safety defined as incidence of device related MAE, defined as amputations or re-interventions (surgical or endovascular)

IPD SHARING:
Plan to Share IPD: No